CLINICAL TRIAL: NCT04329481
Title: The Effect of Mycobiome Supplementation on Gastrointestinal Symptoms in IBD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, PI, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TASMC-17-0643-TLV
Record Dates: First submitted 2020-03-29; First posted 2020-04-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Ulcerative Colitis; Crohn Disease; Inflammatory Bowel Diseases
Keywords: ulcerative colitis; crhon's disease; inflammatory bowel disease; mycobiome
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: The crossover study design is suitable for the aims of this study given that Crhon disease (CD) and ulcerative colitis (UC) patients are both chronic conditions. The treatment investigated is hypothesized to effect patient's symptoms and consequent quality of life.
  Patients will be screened and randomly allocated to be treated with 'Mycodigest' supplementation or placebo for 8 weeks.
  Between the two interventional periods, all participants will undergo a wash-out period of 2 weeks in order to address the potential carryover effect of the first period. As the microbiome is known change rapidly, we assume that this time period will be suitable for minimizing the potential carryover effect of the first period intervention
Who Masked: Participant, Care Provider, Investigator
Masking Description: "Mycodigest" supplementation and placebo will be manufactured by 'Mycolivia Medicinal Mushrooms' LTD, to be identical in size, shape and color.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mycodigest supplement (Active Comparator): "Mycodigest" is a dietary supplement which consists of traditional medicinal mushrooms, as essences and grounded powder. These include Shiitake, Maitake, Trametes Coriolus Versicolor, Agaricus.
  Compliance to treatment will be considered as taking 80% of supplement/placebo treatment, and will be monitored by telephone calls and emails to patients during the study phase, and by counting the pills which were not taken at the end of the trial.
  Treatment with "Mycodigest" supplement will initiate with 2 pills/day for 7 days, and gradually rise to 4 pills/day for 7 days, 6 pills/day for 42 days. Thus, the full dose of the treatment will be administered for 6 weeks.
  Interventions: Dietary Supplement: Mycodigest supplement
- placebo (Placebo Comparator): will be be identical in size, shape and color to "Mycodigest" Treatment with "Mycodigest" placebo will initiate with 2 pills/day for 7 days, and gradually rise to 4 pills/day for 7 days, 6 pills/day for 42 days. Thus, the full dose of the treatment will be administered for 6 weeks.
  Interventions: Dietary Supplement: Mycodigest supplement

INTERVENTIONS:
Dietary Supplement: Mycodigest supplement — Mycodigest" is a dietary supplement which consists of traditional medicinal mushrooms, as essences and grounded powder

SUMMARY:
Studies demonstrated that fungi have a complex, multifaceted role in the gastrointestinal tract and are active participants in directly influencing health and disease through fungal-bacterial, fungal-fungal and fungal-host interactions.

Fungi have been linked with a number of gastrointestinal diseases including IBD, However, the exact role of fungal colonization in the pathophysiology of "IBD" (inflammatory bowel diseases) is not precisely defined.

Aim to evaluate the impact of "Mycodigest" supplementation to IBD patients on: Clinical response and remission rates , Quality of life, Inflammatory markers, Fecal microbiome

DETAILED DESCRIPTION:
Inflammatory bowel diseases ("IBD") are a group of chronic immune-mediated diseases with typical onset during young adulthood and a lifelong course characterized by periods of remission and relapse. IBDs involving two main clinical forms- Crohn's disease ("CD") and ulcerative colitis (UC). CD can affect any part of the gastrointestinal tract with the frequent presentation of abdominal pain, fever, weight loss, and clinical signs of bowel obstruction or diarrhea. In comparison,ulcerative colitis ("UC), in which Inflammation is restricted to the mucosal surface of the colon, manifesting as continuous areas of inflammation, ulceration, edema and hemorrhage. Usually both conditions are chronic, though ulcerative colitis is curable by surgical removal of the colon. Apart from this, there is no cure for IBD. both CD and UC can be treated with medications that induce and maintain remission. Pharmaceutical treatment includes five major categories, namely anti-inflammatory drugs, immune suppressants, biologic agents, antibiotics, and drugs for symptomatic relief. Choice of therapy depends largely on the severity of disease, and may also be influenced by such factors as disease location, side effects and adverse events, as well as cost. The etiology of IBD has been extensively studied in the past few decades however, the pathogenesis is not well understood. several factors that make a major contribution to disease pathogenesis have been identified and distinct to three categories: genetic factors, environmental factors including breast feeding, diet, smoking, drugs etc and microbial factors, producing sustained inflammation supported by altered mucosal barrier and defects in immune system. This combination of features has made IBD both an appropriate and a high-priority platform for translatable research in host-microbiome interactions.

Studies demonstrated that fungi have a complex, multifaceted role in the gastrointestinal tract and are active participants in directly influencing health and disease through fungal-bacterial, fungal-fungal and fungal-host interactions.

Fungi have been linked with a number of gastrointestinal diseases including IBD, However, the exact role of fungal colonization in the pathophysiology of IBD is not precisely defined. study have shown that the diversity and composition of the fungal communities varies in IBD.

A study that characterized the fungal microbiota in the intestinal mucosa and feces in patients with CD found that the fungal richness significantly elevated in the inflamed mucosa compared with the noninflamed mucosa.

This suggests that in IBD, the mycobiome and microbiome have a mutual influence on each other. Pointing to the role of the bacteria and microbial dysbiosis in IBD.

Aims

To evaluate the impact of "Mycodigest" supplementation to inflammatory bowel disease (IBD) patients on:

1. Clinical response and remission rates
2. Quality of life
3. Inflammatory markers
4. Fecal microbiome composition and diversity

ELIGIBILITY:
Inclusion Criteria:

1. Clinically stable patients, constant medicinal regimen throughout the study period. Refractory to mesalamine at least 6 weeks, or steroids at least 2 week, or immunomodulator at least 12 weeks or biologics at least 12 weeks therapy, medical cannabis at least 2 weeks before the study.
2. Patients will be included if they have mild to moderate disease defines as:

   2.1 CD patients will be included if their symptoms score 4<between <16 on the Harvey-Bradshaw index (HBI) score, or HBI < 4 and calprotectin >250 2.2 UC patients will be included if their symptoms score >3between <11 on the SCCAI score, or UC patients with SCCAI <3 and calprotectin >250
3. Patients who agreed to refrain from over the counter (OTC) medications for lower GI symptoms and dietary supplements or other foods containing fermented live bacteria throughout the study period

Exclusion Criteria:

1. Any proven current infection such as Clostridium difficile infection , positive stool culture, or parasites, in cases when a patient complains of diarrhea and have not preformed those tests in the past 6 months
2. Antibiotic use during participation in the study
3. Change in medication regimen before study initiation (see inclusion criteria 2) or during the study
4. Inability to sign informed consent and complete study protocol
5. Pregnancy
6. Subjects with chronic conditions such as cancer, organ transplant subjects, advanced kidney or liver disease, systemic inflammatory conditions other than IBD.
7. Patients with ileostomy, pouch or short bowel

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-12 (Actual); Primary Completion 2022-06-12 (Estimated); Study Completion 2024-06-12 (Estimated)

PRIMARY OUTCOMES:
efficacy of "Mycodigest" supplementation to inflammatory bowel disease (IBD) patients on clinical response and remission rates | week 8
  During the study follow-up remission will be determined by an HBI score <4 for CD and a SCCAI score <2 for UC
efficacy of "Mycodigest" supplementation to inflammatory bowel disease (IBD) patients on clinical response and remission rates | week 18
  During the study follow-up remission will be determined by an HBI score <4 for CD and a SCCAI score <2 for UC
efficacy of "Mycodigest" supplementation to inflammatory bowel disease (IBD) patients on inflammatory markers | week 8
  During the study follow-up inflammatory markers will be determined by CRP concentration <5 mg/L, fecal calprotectin concentration <250 μg/g for both.
efficacy of "Mycodigest" supplementation to inflammatory bowel disease (IBD) patients on inflammatory markers | week 18
  During the study follow-up inflammation markers will be determined by CRP concentration <5 mg/L, fecal calprotectin concentration <250 μg/g for both.

SECONDARY OUTCOMES:
efficacy of "Mycodigest" supplementation to inflammatory bowel disease (IBD) patients on quality of life | week 8
  During the study quality of life will be assessed by filling a quality of life questionnaire that will be compared between the baseline and week 8. The is no scale to the questionnaire.
efficacy of "Mycodigest" supplementation to inflammatory bowel disease (IBD) patients on quality of life | week 18
  During the study quality of life will be assessed by filling a quality of life questionnaire that will be compared between the baseline and week 18. The is no scale to the questionnaire.
effect of "Mycodigest" supplementation to inflammatory bowel disease (IBD) patients on 4. Fecal microbiome composition and diversity | week 8
  Fecal microbiome composition and diversity will be assessed by- DNA will be extracted from the stool using PowerLyzer PowerSoil DNA isolation kit (MoBio) for characterizing the microbial composition. DNA extraction will be followed by PCR amplification of the V3-V4 regions of the bacterial 16S rRNA gene, using 515F/806R primers. Last, 500 bp paired-end sequencing will be performed on an Illumina MiSeq. The collected data will be analyzed using the QIIME pipeline. Following the pipeline we will filter and normalize the data by applying a bottom threshold of 0.002 relative abundance to all values under detection level (0 to 0.002) and only taxa. For beta-diversity, unweighted unifrac measurements will be plotted according to the first two principal coordinates based on 9,000 reads per sample.
effect of "Mycodigest" supplementation to inflammatory bowel disease (IBD) patients on 4. Fecal microbiome composition and diversity | week 18
  Fecal microbiome composition and diversity will be assessed by- DNA will be extracted from the stool using PowerLyzer PowerSoil DNA isolation kit (MoBio) for characterizing the microbial composition. DNA extraction will be followed by PCR amplification of the V3-V4 regions of the bacterial 16S rRNA gene, using 515F/806R primers. Last, 500 bp paired-end sequencing will be performed on an Illumina MiSeq. The collected data will be analyzed using the QIIME pipeline. Following the pipeline we will filter and normalize the data by applying a bottom threshold of 0.002 relative abundance to all values under detection level (0 to 0.002) and only taxa. For beta-diversity, unweighted unifrac measurements will be plotted according to the first two principal coordinates based on 9,000 reads per sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroentherology, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No